CLINICAL TRIAL: NCT03963102
Title: A Study to Investigate the Effect of Different Durations of Ameluz Application on Response to Treatment of Acral Actinic Keratoses
Brief Title: Duration of Ameluz Application in Acral Actinic Keratoses Response
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of appropriate personnel. Dr Xie abroad on other research, current PI Dr John Frewen not at main centre, no other available PI identified. Study suspended.
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PDT AK v1
Record Dates: First submitted 2019-03-19; First posted 2019-05-24 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Actinic Keratoses; Photodamaged Skin
Keywords: photodynamic therapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: Randomised control study, prospective, assessor blinded.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor is blinded to whether the patient is in the control or trial group when assessing the primary outcome at 3 months. There will be an additional member of staff present to ensure blinding is not revealed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group 3 hours (Active Comparator): Application of Ameluz for 3 hours.
  Interventions: Drug: Ameluz
- Trial Group 4 hours (Experimental): Application of Ameluz for 4 hours.
  Interventions: Drug: Ameluz

INTERVENTIONS:
Drug: Ameluz — Leaving on the gel for 4 hours rather than the standard 3 hours.

SUMMARY:
A phase IV study of a single topical application of ALA for 3 hours or 4 hours to AK on acral sites (hands, feet, arms and legs), and subsequent measurement of clinical efficacy with corresponding PpIX fluorescence imaging.

DETAILED DESCRIPTION:
Photodynamic therapy (PDT) is a relatively new treatment for skin cancer and sun-damaged skin, which may turn cancerous or pre-cancerous. PDT treatment consists of applying a gel containing aminolevulinic acid hydrochloride (licensed for clinical use as Ameluz®) to the abnormal area. Inside the diseased cells this gel is changed over a few hours into a light-sensitive chemical (photosensitiser) that reacts with light. The photosensitiser is inactive by itself. A red light is then shone on to the lesion; this reacts with the photosensitiser and destroys the abnormal cells. Only the treated area will be affected and inflamed. The area will be cured in most cases after the inflammation clears.

Actinic keratosis (AK) is a type of pre-cancerous lesion caused by sun damage. If left, they can progress to become skin cancer. These can be treated in different ways, with different topical creams, liquid nitrogen or PDT. Some lesions may have reoccurred after topical creams, patients also have unacceptable amount of inflammation or the lesion involve too large an area. Liquid nitrogen is as good as PDT in treating AKs, however have been reported to leave a less good cosmetic result.

PDT is a licensed treatment for AK. However, PDT has been shown to be less effective for AKs on certain areas such as hands and feet. Further understanding of the build-up of the photosensitiser may enable better cure rates at these body parts, enabling more patients to benefit from PDT.

The proposed theory is that a longer application of the Ameluz gel will increase the amount of photosensitiser, which accumulates in the treated areas, and thus increase the amount of damage to cells, and mean that more patients have a successful treatment.

The aim of this study is to investigate whether applying the Ameluz gel for 4 hours (trial group) rather than 3 hours (control group) will improve treatment success rates in AK lesions on hands, feet, arms and legs. The information gained from this study may result in better treatment design of PDT for AK.

To do this the investigators plan to apply Ameluz® gel to AK lesions for either the standard 3 hours or the currently unlicensed 4 hours. The investigators will then measure the amount of that has changed into the photosensitiser, using a special digital camera. This camera device is not invasive and does not have any side effects. Some patients may have multiple AK lesions on multiple sites; the investigator aim to treat all these in the same manner due to practicality, and will record data for these lesions as well.

The investigator will record if patients report any associated pain during light delivery, as well as the temperature of the lesion during treatment. Some patients opt to have an external cooling system or water spray during the light treatment, but in order to standardise treatment during the trial this will not be used. The investigator will however give patients the option of taking paracetamol themselves prior to the treatment. A dermatology doctor will then review the patients at three months following treatment to see if their AK has been cured, and receive further treatment if needed.

The pathway is the same as standard PDT treatment and does not involve an extra visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has given written informed consent.
2. Males and females > 18 years.
3. AK lesions on arms, hands, legs or feet that are practical to treat with PDT.

Exclusion Criteria:

1. Lesions with a clinical diagnosis of Bowen's disease, superficial, morphoeic or nodular basal cell carcinoma, squamous cell carcinoma, or melanoma as they are not the types of lesions required for investigation.
2. Any disease which is caused or exacerbated by light, including systemic lupus erythematosus, porphyria, actinic reticuloid or xeroderma pigmentosum. Part of the clinical study will be the use of light-imaging system so any condition, which is sensitive to such instruments, will be excluded.
3. Males or females of childbearing potential, who are not practicing adequate contraceptive precaution. Female patients should practice strict birth control (oestrogen-containing oral contraceptives or an IUD) throughout the trial. Only post-menopausal women (12 months or more with no menses) and women who have had a hysterectomy are exempt from the requirements to use birth control. Male patients should also use adequate contraception for the duration of the trial.
4. Pregnant or lactating females
5. Treatment in the previous 45 days with any cryotherapy, topical treatments for AK, experimental compound, an iron chelating agent, radiotherapy, chemotherapy or with any light activated therapy or any other medication, which may render the patient light sensitive (e.g. PUVA).
6. Photodynamic therapy treatment in the previous 90 days.
7. Co-existing ophthalmic disease likely to require slit lamp examination within 30 days of PDT treatment.
8. Known allergies to porphyrins, peanut, soya or excipients.
9. Patients not able to comply with study requirements.
10. Patients on immunosuppression medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The odds of full clearance of individual lesions in the intervention and control groups will be compared (reported as an odds ratio with 95%CLs). | 3 months
  Clinical outcome at 3 months of the treated AK lesions on acral sites

SECONDARY OUTCOMES:
Clearance of lesions on other body sites | 3 months
  The odds of full clearance of any non-acral individual lesions in the intervention and control groups will be compared (reported as an odds ratio with 95%CLs). Lesions will be either cleared or not cleared.
Pain Score | 1 week
  The mean of pain levels as measure by the Visual Analogue Scale with standard deviation will be provided between treatment arms.
Photobleaching | After data collection is completed, during analysis phase, expected at 12 months.
  Photobleaching will be calculated as the difference in fluorescence score before and after light treatment (change score). This is measured using the Dyaderm Fluroscence imaging system.
PpIX accumulation fluorescence | After data collection is completed, during analysis phase, expected at 12 months.
  PpIX accumulation over time (3 measurements for each lesion) will be presented graphically, grouped by participant and lesion type (acral and non-acral). The accumulation score is the PpIX fluroscence measured before light treatment.
  The fluorescence before light treatment will be compared between intervention and control groups with a random effects model. The analysis will be adjusted for baseline fluorescence, grade of lesion, and location of lesion. A change score analysis will be carried out for comparison.
PpIX dissipation fluorescence | After data collection is completed, during analysis phase, expected at 12 months.
  PpIX dissipation over time (3 measurements for each lesion) will be presented graphically, grouped by participant and lesion type (acral and non-acral). The dissipation score is the PpIX fluroscence measured after light treatment.
  The fluorescence after light treatment will be compared between intervention and control groups with a random effects model. The analysis will be adjusted for baseline fluorescence, grade of lesion, and location of lesion. A change score analysis will be carried out for comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Cornwall Hospital, Truro, Cornwall, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Please contact study coordinators to see if non-patient identifiable information can be release.